CLINICAL TRIAL: NCT00618293
Title: Phase 2 Study in Evaluation of the Efficacy and Safety of Haemate HS in This Clinical Setting (Patients With Severe Bleeding Undergoing Valve Replacement Due to Aortic Stenosis)
Brief Title: Haemate HS in Patients With Severe Bleeding Undergoing Valve Replacement Due to Aortic Stenosis
Acronym: HAVAS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patient met the criteria for inclusion in the study.
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Heinrich-Heine University, represented by Principal investigator Prof. Feindt, Department of Hemostasis and Transfusion Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BI8021_5101
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Blood Loss, Surgical
Keywords: intraoperative bleeding; aortic-valve replacement; aortic stenosis; Von Willebrand; HEAMATE
MeSH Terms: conditions — Blood Loss, Surgical; Aortic Valve Stenosis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): intravenous infusion of Haemate (dosage dependent on body weight)
  Interventions: Drug: Haemate HS
- 2 (Placebo Comparator): intravenous infusion of 0.9% NaCl solution
  Interventions: Other: NaCl-solution

INTERVENTIONS:
Drug: Haemate HS — intravenous infusion of Haemate (dosage dependent on body weight)
  Arms: 1
Other: NaCl-solution — intravenous infusion of 0.9%NaCl-Solution
  Arms: 2

SUMMARY:
Evaluation of efficacy by determination of transfusion requirements and safety by determination of adverse events in administration of Von Willebrand factor concentrate F VIII (Haemate).

ELIGIBILITY:
Inclusion Criteria:

* patients with isolated valvular aortic stenosis or combined aortic-valve defect with prevailing stenosis with severe bleeding during aortic-valve replacement
* Caucasian
* written informed consent (Classification of bleeding as "normal", "moderate" or "excessive" by the surgeon.Classification as excessive leads to recruitment)

Exclusion Criteria:

* active endocarditis
* history suggestive for inherited oe acquired bleeding disorder
* concomitant coronary heart disease
* agents impairing platelet function up to 14 days before surgery
* Pregnancy
* inherited platelet function
* known intolerance against HAEMATE HS
* previous thromboembolic complications
* Hepatitis B, C or HIV infection
* previous chemotherapy
* emergency surgery within the last 7 days
* weight < 50 kg and > 100 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Estimated); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
intra- and postoperative transfusion requirements of packed red cells, platelet concentrates and fresh frozen plasma according to defined transfusion thresholds | begin of surgery and 48h after administration of medication

SECONDARY OUTCOMES:
Assessment of adverse events and viral safety | 1.perioperative 2. during hospital admission 3. within 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feindt, Prof. Dr. med., Principal Investigator — Klinik für Kardiovaskuläre Chirurgie
Locations (1):
- Klinik für Kardiovaskuläre Chirurgie, Düsseldorf, Germany